CLINICAL TRIAL: NCT05026723
Title: Food as Medicine for HIV: A Randomized Trial of Medically Tailored Meals and Lifestyle Intervention
Brief Title: Food as Medicine for HIV and Diabetes
Acronym: FAME-H
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Community Servings (Other); Massachusetts General Hospital (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-3509; R01DK127365 (NIH)
Record Dates: First submitted 2021-08-23; First posted 2021-08-30 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2; HIV Infections; PreDiabetes
Keywords: Food Insecurity; Socioeconomic Factors; Lifestyle Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; HIV Infections; Prediabetic State | interventions — myotubularin

STUDY DESIGN:
Intervention Model Description: Participants will be assigned in 1:1 ratio to one of two intervention arms
Who Masked: Outcomes Assessor
Masking Description: Owing to the nature of the intervention, participants, providers, and many study staff will know to which group individual participants have been randomized. However, efforts will be made to keep the study statistician and outcome assessors blinded to randomization group during the course of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medically Tailored Meal (MTM) + Intensive Lifestyle Intervention (ILI) (Experimental): The Medically Tailored Meal (MTM) + Intensive Lifestyle Intervention (ILI) consists of weekly home meal delivery; an explanation of the medical tailoring of the meals; and a 20-session telephone lifestyle intervention change program designed to complement the period of meal delivery and prepare for the period after meal delivery with behavioral and skill-building approaches to sustain the benefit of the intervention.
  Interventions: Behavioral: MTM + ILI
- Standard MTM (Active Comparator): The Standard Medically Tailored Meal (MTM) intervention (ILI) consists of weekly home meal delivery; an explanation of the medical tailoring of the meals; and an initial consultation with a dietitian.
  Interventions: Behavioral: Standard MTM

INTERVENTIONS:
Behavioral: MTM + ILI — Weekly home meal delivery; an explanation of the medical tailoring of the meals; and a 20-session telephone lifestyle intervention change program
  Arms: Medically Tailored Meal (MTM) + Intensive Lifestyle Intervention (ILI)
Behavioral: Standard MTM — Weekly home meal delivery; an explanation of the medical tailoring of the meals; and an initial consultation with a dietitian
  Arms: Standard MTM

SUMMARY:
This is a single-site, open-label, Phase II, community-based randomized controlled explanatory trial to test the efficacy of a medically tailored meal + intensive lifestyle intervention (MTM + ILI) intervention for adults with food insecurity, HIV, and T2DM or high risk of T2DM, compared with a group that receives usual MTM.

DETAILED DESCRIPTION:
In contemporary practice for people with HIV, type 2 diabetes mellitus (T2DM) has become an important comorbidity. T2DM is 1.5 times more common in people with HIV than the general population. Among those with T2DM, people with HIV have greater risk for weight gain, lower diet quality, and higher hemoglobin A1c. All of this puts people with HIV and T2DM at substantial risk for complications, including chronic kidney disease, cardiovascular disease, and premature mortality. Food insecurity, "lack of access to enough food for an active, healthy life", is a major contributor to this risk. Food insecurity is 2 to 3 times more common among people with HIV than the general population. Food insecurity is associated with both worse T2DM control and more T2DM complications.

Medically tailored meal home delivery programs relieve food insecurity for people with HIV. Medically tailored meals emerged to treat food insecurity among those with AIDS in the 1990's. Medically tailored meal programs deliver fully prepared meals, tailored by a registered dietitian to an individual's medical needs. Although HIV care has changed, medically tailored meal interventions for people with HIV have not kept pace. Most medically tailored meal programs do not provide the intensive lifestyle intervention needed to counter the health threats seen in modern HIV care. These threats include the metabolic effects of anti-retroviral medications, chronic inflammation, aging, and obesogenic environments. For these reasons, it is critical to test new models of medically tailored meal for people with HIV.

The investigators has developed a medically tailored meal intervention that combines meal delivery with an evidence-based lifestyle intervention designed to improve weight loss and diabetes self-management. The goal for this project is to test whether this medically tailored meal intervention can lead to improvements in weight, hemoglobin A1c, and in patient-reported outcomes such as food insecurity, quality of life, and diabetes distress, compared with a standard medically tailored meal intervention.

Thus, the investigators propose a randomized comparative effectiveness trial to assess a community-based medically tailored meals intervention (n=200). It will be conducted among diverse participants with HIV and T2DM or high risk for T2DM, referred for medically tailored meals. Adults with hemoglobin A1c less than 12.0%, and BMI ≥ 23 kg/m^2 will be enrolled and randomly assigned to intervention or standard medically tailored meals. The intervention group will receive meal delivery and intensive lifestyle intervention for 12 months, while the comparison group will receive meal delivery along with standard nutrition education for 12 months. Outcomes will be assessed at 6, 12, and 18 months. The primary outcome is weight at 6 months. Secondary outcomes include hemoglobin a1c, food security, quality of life, and diabetes distress.

ELIGIBILITY:
Inclusion Criteria

* Male or female
* Diagnosis of HIV
* Diagnosis of Type 2 Diabetes Mellitus or high risk for type 2 diabetes mellitus, defined as meeting CDC eligibility criteria for the diabetes prevention program. Specifically, an individual without a diagnosis of T2DM must 1) have had a blood test result in the prediabetes range within the past year (Hemoglobin A1C: 5.7-6.4% OR Fasting plasma glucose: 100-125 mg/dL OR Two-hour plasma glucose [after a 75 g glucose load]: 140-199 mg/dL), 2) Have been previously diagnosed with gestational diabetes, OR 3) have a high-risk result (score of 5 or higher) on the Prediabetes Risk Test (https://www.cdc.gov/prediabetes/pdf/Prediabetes-Risk-Test-Final.pdf)
* Experiencing food insecurity as indicated by 2-item Hunger Vital Sign
* English speaking
* Aged ≥18 years
* BMI ≥ 23 kg/m2
* No plans to move from the area for at least 1 year
* Free living to the extent that participant has control over dietary intake
* Willing and able to provide written informed consent and participate in all study activities

Exclusion Criteria:

* Participant in diabetes, nutrition, or weight research intervention in last 12 months
* Current AIDS defining illness
* Another family member or household member is a study participant. Only one member of each household may take part in this study.
* Considering bariatric surgery in the next year or prior bariatric surgery in the past 2 years
* Lack of safe, stable residence and ability to store meals
* Lack of telephone
* Pregnancy/breastfeeding or intended pregnancy in the next year
* History of malignancy, other than non-melanoma skin cancer, unless surgically or medically cured > 5 years ago or in remission. Patients with localized prostate and breast cancer diagnosed during the course of routine screening will not be excluded.
* Advanced kidney disease (estimated creatinine clearance < 30 ml/min)
* Known drug or alcohol misuse in the past 6 months
* Known psychosis or major psychiatric illness that prevents participation with study activities
* Intermittent use of medications (e.g., oral or intravenous glucocorticoids) that are likely to affect blood sugar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Bodyweight at Month 6 | 6 months
  Bodyweight measured in Kg

SECONDARY OUTCOMES:
Bodyweight at Month 12 | 12 months
  Bodyweight measured in Kg
Bodyweight at Month 18 | 18 months
  Bodyweight measured in Kg
Hemoglobin A1c at Month 6 | 6 months
  Hemoglobin A1c Level
Hemoglobin A1c at Month 12 | 12 months
  Hemoglobin A1c Level
Hemoglobin A1c at Month 18 | 18 months
  Hemoglobin A1c Level
Health-Related Quality of Life Score as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS)-29 at Month 6 | 6 months
  The PROMIS-29 includes seven health related quality of life domains (Physical Functioning, Anxiety, Depression, Fatigue, Sleep Disturbance, Social Functioning, and Pain), and the pain domain has two subdomains (interference and intensity). Raw scores, except pain intensity, are transformed using the T-score metric based on the item response theory calibrations in which scores have a mean of 50 and standard deviation of 10 for the general population in the US. A higher PROMIS T-score implies more of the concept being measured; i.e., a higher PROMIS score on physical function indicates better functioning, whereas a higher score on depression indicates more severe depressive symptoms. Will report overall score and scores for each domain. From these data will also calculate a PROMIS-Preference (PROPr score) (PROPr scores range from -0.022 (worst) to 1.0 (best)).
Health-Related Quality of Life Score as assessed by PROMIS-29 at Month 12 | 12 months
  The PROMIS-29 includes seven health related quality of life domains (Physical Functioning, Anxiety, Depression, Fatigue, Sleep Disturbance, Social Functioning, and Pain), and the pain domain has two subdomains (interference and intensity). Raw scores, except pain intensity, are transformed using the T-score metric based on the item response theory calibrations in which scores have a mean of 50 and standard deviation of 10 for the general population in the US. A higher PROMIS T-score implies more of the concept being measured; i.e., a higher PROMIS score on physical function indicates better functioning, whereas a higher score on depression indicates more severe depressive symptoms. Will report overall score and scores for each domain. From these data will also calculate a PROMIS-Preference (PROPr score) (PROPr scores range from -0.022 (worst) to 1.0 (best)).
Health-Related Quality of Life Score as assessed by PROMIS-29 at Month 18 | 18 months
  The PROMIS-29 includes seven health related quality of life domains (Physical Functioning, Anxiety, Depression, Fatigue, Sleep Disturbance, Social Functioning, and Pain), and the pain domain has two subdomains (interference and intensity). Raw scores, except pain intensity, are transformed using the T-score metric based on the item response theory calibrations in which scores have a mean of 50 and standard deviation of 10 for the general population in the US. A higher PROMIS T-score implies more of the concept being measured; i.e., a higher PROMIS score on physical function indicates better functioning, whereas a higher score on depression indicates more severe depressive symptoms. Will report overall score and scores for each domain. From these data will also calculate a PROMIS-Preference (PROPr score) (PROPr scores range from -0.022 (worst) to 1.0 (best)).
Depressive Symptom Score at Month 6 | 6 months
  Depressive Symptoms as assessed by PROMIS Short Form (PROMIS SF) v1.0 - Depression 4a. Raw scores are transformed using the T-score metric based on the item response theory calibrations in which scores have a mean of 50 and standard deviation of 10 for the general population in the US. A higher PROMIS T-score implies more of the concept being measured; i.e., a higher PROMIS score on depression indicates more severe depressive symptoms.
Depressive Symptom Score at Month 12 | 12 months
  Depressive Symptoms as assessed by PROMIS SF v1.0 - Depression 4a. Raw scores are transformed using the T-score metric based on the item response theory calibrations in which scores have a mean of 50 and standard deviation of 10 for the general population in the US. A higher PROMIS T-score implies more of the concept being measured; i.e., a higher PROMIS score on depression indicates more severe depressive symptoms.
Depressive Symptom Score at Month 18 | 18 months
  Depressive Symptoms as assessed by PROMIS SF v1.0 - Depression 4a. Raw scores are transformed using the T-score metric based on the item response theory calibrations in which scores have a mean of 50 and standard deviation of 10 for the general population in the US. A higher PROMIS T-score implies more of the concept being measured; i.e., a higher PROMIS score on depression indicates more severe depressive symptoms.
Diabetes Distress Score as assessed by Problem Areas in Diabetes (PAID)-11 at Month 6 | 6 months
  Score ranges from 11-55 with higher scores indicating greater diabetes distress
Diabetes Distress Score as assessed by PAID-11 at Month 12 | 12 months
  Score ranges from 11-55 with higher scores indicating greater diabetes distress
Diabetes Distress Score as assessed by PAID-11 at Month 18 | 18 months
  Score ranges from 11-55 with higher scores indicating greater diabetes distress

OTHER OUTCOMES:
Food Insecurity Score at Month 6 | 6 Months
  Food Insecurity Score. Score ranges from 0-10, with higher scores indicating greater food insecurity.
Food Insecurity Score at Month 12 | 12 Months
  Food Insecurity Score. Score ranges from 0-10, with higher scores indicating greater food insecurity.
Food Insecurity Score at Month 18 | 18 Months
  Food Insecurity Score. Score ranges from 0-10, with higher scores indicating greater food insecurity.
Systolic Blood Pressure at Month 6 | 6 Months
  Systolic blood pressure in mm Hg
Systolic Blood Pressure at Month 12 | 12 Months
  Systolic blood pressure in mm Hg
Systolic Blood Pressure at Month 18 | 18 Months
  Systolic blood pressure in mm Hg
Diastolic Blood Pressure at Month 6 | 6 Months
  Diastolic blood pressure in mm Hg
Diastolic Blood Pressure at Month 12 | 12 Months
  Diastolic blood pressure in mm Hg
Diastolic Blood Pressure at Month 18 | 18 Months
  Diastolic blood pressure in mm Hg
Diet Quality Score at Month 6 | 6 months
  Diet Quality as assessed by Brief Dietary Assessment Scale. This score is comprised of 3 sections (or subscales) used to assess dietary patterns. Subscales are scored independently. The subscales are: Vegetables, Fruit, Whole Grains, and Beans subscale (range 0 - 20), Drinks, Desserts, Snacks, Eating Out, and Salt subscale (range 0- 20), and Fish, Meat, Poultry, Dairy, and Eggs subscale (range 0-10): Total score equals the sum of the 3 subscales. For subscales and total score, higher scores indicates better diet quality.
Diet Quality Score at Month 12 | 12 months
  Diet Quality as assessed by Brief Dietary Assessment Scale. This score is comprised of 3 sections (or subscales) used to assess dietary patterns. Subscales are scored independently. The subscales are: Vegetables, Fruit, Whole Grains, and Beans subscale (range 0 - 20), Drinks, Desserts, Snacks, Eating Out, and Salt subscale (range 0- 20), and Fish, Meat, Poultry, Dairy, and Eggs subscale (range 0-10): Total score equals the sum of the 3 subscales. For subscales and total score, higher scores indicates better diet quality.
Diet Quality Score at Month 18 | 18 months
  Diet Quality as assessed by Brief Dietary Assessment Scale. This score is comprised of 3 sections (or subscales) used to assess dietary patterns. Subscales are scored independently. The subscales are: Vegetables, Fruit, Whole Grains, and Beans subscale (range 0 - 20), Drinks, Desserts, Snacks, Eating Out, and Salt subscale (range 0- 20), and Fish, Meat, Poultry, Dairy, and Eggs subscale (range 0-10): Total score equals the sum of the 3 subscales. For subscales and total score, higher scores indicates better diet quality.
Cost-Related Medication Underuse at Month 6 | 6 months
  Any affirmative response to cost-related medication underuse items
Cost-Related Medication Underuse at Month 12 | 12 months
  Any affirmative response to cost-related medication underuse items
Cost-Related Medication Underuse at Month 18 | 18 months
  Any affirmative response to cost-related medication underuse items
Adherence to Refills and Medications Scale-Diabetes (ARMS-D) Medication Adherence Score at Month 6 | 6 months
  Medication Adherence as assessed by 7-item ARMS-D scale. Scores range from 7 to 28, with higher scores indicating more problems with adherence.
ARMS-D Medication Adherence Score at Month 12 | 12 months
  Medication Adherence as assessed by 7-item ARMS-D scale. Scores range from 7 to 28, with higher scores indicating more problems with adherence.
ARMS-D Medication Adherence Score at Month 18 | 18 months
  Medication Adherence as assessed by 7-item ARMS-D scale. Scores range from 7 to 28, with higher scores indicating more problems with adherence.
Diabetes Self-Care Activities Medication Adherence Score at Month 6 | 6 months
  Medication Adherence as assessed by 1-item summary of diabetes self-care activities measure. Scores range from 0-7 with higher scores indicating better adherence.
Diabetes Self-Care Activities Medication Adherence Score at Month 12 | 12 months
  Medication Adherence as assessed by 1-item summary of diabetes self-care activities measure. Scores range from 0-7 with higher scores indicating better adherence.
Diabetes Self-Care Activities Medication Adherence Score at Month 18 | 18 months
  Medication Adherence as assessed by 1-item summary of diabetes self-care activities measure. Scores range from 0-7 with higher scores indicating better adherence.
Diet Self-Efficacy Score at Month 6 | 6 months
  Diet Self-Efficacy as assessed by cardiac diet self-efficacy scale. Scores range from 16 to 80 with higher scores indicating greater self-efficacy.
Diet Self-Efficacy Score at Month 12 | 12 months
  Diet Self-Efficacy as assessed by cardiac diet self-efficacy scale. Scores range from 16 to 80 with higher scores indicating greater self-efficacy.
Diet Self-Efficacy Score at Month 18 | 18 months
  Diet Self-Efficacy as assessed by cardiac diet self-efficacy scale. Scores range from 16 to 80 with higher scores indicating greater self-efficacy.
Perceived Diabetes Self-Management Self-Efficacy Score at Month 6 | 6 months
  Diabetes Self-Efficacy as assessed by Perceived Diabetes Self-Management Scale. Scores range from 8 to 40 with higher scores indicating greater self-efficacy
Perceived Diabetes Self-Management Self-Efficacy Score at Month 12 | 12 months
  Diabetes Self-Efficacy as assessed by Perceived Diabetes Self-Management Scale. Scores range from 8 to 40 with higher scores indicating greater self-efficacy
Perceived Diabetes Self-Management Self-Efficacy Score at Month 18 | 18 months
  Diabetes Self-Efficacy as assessed by Perceived Diabetes Self-Management Scale. Scores range from 8 to 40 with higher scores indicating greater self-efficacy
Stress Score at 6 months | 6 months
  Stress as assessed by perceived stress scale. Scores range from 0 to 40 with higher scores indicating higher perceived stress.
Stress Score at 12 months | 12 months
  Stress as assessed by perceived stress scale. Scores range from 0 to 40 with higher scores indicating higher perceived stress.
Stress Score at 18 months | 18 months
  Stress as assessed by perceived stress scale. Scores range from 0 to 40 with higher scores indicating higher perceived stress.
Food/Medication Trade-offs at Month 6 | 6 months
  Single item-indicators of trading off medication for food or food for medication. An affirmative response indicates the presence of a trade-off.
Food/Medication Trade-offs at Month 12 | 12 months
  Single item-indicators of trading off medication for food or food for medication. An affirmative response indicates the presence of a trade-off.
Food/Medication Trade-offs at Month 18 | 18 months
  Single item-indicators of trading off medication for food or food for medication. An affirmative response indicates the presence of a trade-off.
Cluster of Differentiation 4 (CD4+) Count at Month 6 | 6 Months
  CD4+ Count
Self-Reported CD4+ Count at Month 6 | 6 Months
  Self-Reported CD4+ Count
Self-Reported CD4+ Count at Month 12 | 12 Months
  Self-Reported CD4+ Count
Self-Reported CD4+ Count at Month 18 | 18 Months
  Self-Reported CD4+ Count
HIV Viral Load at Month 6 | 6 Months
  HIV Viral Load
Self-Reported HIV Viral Load at Month 6 | 6 Months
  Self-Reported HIV Viral Load
Self-Reported HIV Viral Load at Month 12 | 12 Months
  Self-Reported HIV Viral Load
Self-Reported HIV Viral Load at Month 18 | 18 Months
  Self-Reported HIV Viral Load
C-Reactive Protein (CRP) at Month 6 | 6 months
  C-Reactive Protein

CONTACTS AND LOCATIONS:
Overall Officials: Seth A Berkowitz, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that can be deidentified without risk of confidentiality breach will shared upon written request made to study investigators. In addition, all NIH policies regarding data sharing will be followed. Deidentified individual data that supports the results will be shared provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill (UNC).
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Unless preempted by NIH policy, data will become available 12 months after publication of main findings, and be available for 60 months.
Access Criteria: Unless otherwise required by NIH policy, ability to deidentify data, plan for secure storage of data and agreement to protect participant privacy, and relevant research question, to be assessed by study investigators.